CLINICAL TRIAL: NCT05854511
Title: Pharmacokinetics, Safety, Efficacy and Acceptability Study of Daclatasvir/Sofosbuvir in Children Weighing 14-35 Kilograms With Chronic Hepatitis C Virus Infection
Brief Title: Pharmacokinetics, Safety, Efficacy and Acceptability of Daclatasvir Plus Sofosbuvir in HCV-infected Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Manal Hamdy El-Sayed, Professor of Pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P04a / 2022
Record Dates: First submitted 2022-08-21; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: HCV
Keywords: Daclatasvir; Sofosbuvir; Children; HCV; Pharmacokinetics; Safety; Efficacy; Acceptability
MeSH Terms: interventions — Sofosbuvir; Tablets; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daclatasvir Plus Sofosbuvir (Experimental): treatment-naïve children infected with chronic HCV will be stratified according to weight
  1. Children weighing 14 <17 Kg
  2. Children weighting 17<35 Kg
  Interventions: Drug: Sofosbuvir 200 MG Oral Tablet plus Daclatasvir 30 mg Oral tablets

INTERVENTIONS:
Drug: Sofosbuvir 200 MG Oral Tablet plus Daclatasvir 30 mg Oral tablets — Daclatasvir 30 mg orally once daily plus Sofosbuvir at a dose of 200 mg (2x 100 mg tablets) orally once daily for 12 weeks.
  Other Names: Daklinza; Sovaldi

SUMMARY:
This is an interventional, single center, single arm clinical trial to assess the pharmacokinetics, safety, efficacy, and acceptability of daclatasvir plus sofosbuvir in treatment-naïve children weighing between 14 and 35 kg with chronic HCV GT 1-6 infection.

DETAILED DESCRIPTION:
This is an interventional, single center, single arm clinical trial to assess the pharmacokinetics, safety, efficacy, and acceptability of daclatasvir plus sofosbuvir in treatment-naïve, children weighing between 14 and 35 kg with chronic HCV GT 1-6 infection.

All enrolled patients will receive daclatasvir 30 mg orally once daily plus sofosbuvir at a dose of 200 mg (2x 100 mg tablets) orally once daily for 12 weeks.

Patients will be followed closely for disease progression and any hypersensitivity or adverse reactions due to therapy. Laboratory values to be monitored at baseline are serum creatinine, bilirubin, Aspartate transaminase (AST), Alanine transaminase (ALT), viral load (VL).

patients will be recruited in each of two weight bands (14 to < 17 kg and 17 to 35 kg). The study is mainly powered for non-compartmental pharmacokinetics determination of DCV, SOF and GS-331007. Patient recruitment will be done at Ain Shams university hospitals, Egypt. The study be will conducted after approval by the corresponding research ethical committee and obtaining an informed consent from the parents or the legal guardians, and -whenever applicable- an assent from the patients.

Total number of visits is 7 for patients who will complete the study, a screening visits, at the first day of therapy, at weeks 1, 4, 8, 12 and 24 after starting daclatasvir plus sofosbuvir. Patients who will complete their treatment schedule will come after 12 weeks for assessment of SVR. Duration of follow up will be 6 months from treatment initiation in addition to screening period (2-4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Children more than 3 years of age and weighing 14-35kg
* Infected with HCV genotypes 1-6
* Treatment Naïve HCV-infected children
* Signing a written consent form by the parent or the legal guardian, and -whenever applicable- an assent by the patient
* Screening laboratory values within predefined thresholds:

  1. Absolute neutrophil count ≥ 1,500/mm3
  2. Platelets > 50,000 cells/mm3
  3. Albumin > 3.5 mg/dL
  4. Prothrombin Time PT < 4 sec above control Or International Normalized Ratio INR <1.7 3
  5. Random blood glucose level within normal range (> 70 mg/dL and < 200 mg/dL)
  6. Serum creatinine < 1.5 mg/dL

Exclusion Criteria:

* Co-infection with HIV, acute hepatitis A virus, or hepatitis B virus
* Clinical hepatic decompensation, i.e., Child-Turcotte-Pugh CTP class B or C (i.e., jaundice, ascites, encephalopathy, or variceal hemorrhage)
* Renal dysfunction, i.e., eGFR < 60 mL/min/1.73 m2 or on regular dialysis as calculated by Schwartz Formula
* Alfa-fetoprotein level > 50 ng/mL
* Chronic liver disease due to a cause other than HCV or Known hypersensitivity to daclatasvir or sofosbuvir.
* History of gastrointestinal disease or gastrointestinal surgical procedure that would impair the absorption of the study drug
* Blood/blood product transfusion within 4 weeks prior to study.
* Systemic corticosteroid administration for more than 2 weeks starting from two weeks before study inclusion and till the end of treatment period (pulmonary/nasal administration is permitted).
* Psychiatric hospitalization, suicide attempt or disability resulting from psychiatric illness within the prior 5 years.
* Ongoing treatment with any medications interacting with daclatasvir/sofosbuvir.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-13 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Daclatasvir | one week
  The plasma concentration of Daclatasvir on day 8 will be used to derive the Pharmacokinetic parameters using the Non-Compartmental analysis (NCA)
Plasma concentration of Sofosbuvir | one week
  The plasma concentration of Daclatasvir on day 8 will be used to derive the Pharmacokinetic parameters using the Non-Compartmental analysis (NCA)

SECONDARY OUTCOMES:
Efficacy of Daclatasvir 30 MG oral tablets and Sofosbuvir 200 MG oral tablets once daily for 12 weeks | 24 weeks
  Efficacy will be assessed via sustained virologic response at 12 weeks after the 12 weeks treatment completion (SVR12)
Safety of Daclatasvir 30 MG oral tablets and Sofosbuvir 200 MG oral tablets once daily for 12 weeks | 24 weeks
  Safety o will be assessed by recording any adverse event occurs in treatment period and 2-4 weeks after the last visit (after week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Manal H. El-Sayed, MD, Principal Investigator — Department of Paediatrics, Faculty of Medicine, Ain Shams University, Cairo, Egypt
Locations (1):
- Faculty of Medicine, Ain-Shams University Research Institute-Clinical Research Centre (MASRI-CRC), Cairo, Egypt